CLINICAL TRIAL: NCT03150641
Title: Maternal Blood Loss With Delayed Cord Clamping During Cesarean Delivery at Term
Brief Title: Delayed Cord Clamping at Term Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAR2937
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Maternal Blood Loss; Cesarean Delivery; Delayed Cord Clamping; Neonatal Health
Keywords: Maternal blood loss; Cesarean delivery; Delayed cord clamping; Neonatal health
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate cord clamping (Other): Umbilical cord clamped within 15 seconds of delivery of baby
  Interventions: Procedure: Umbilical cord clamping
- Delayed cord clamping (Experimental): Umbilical cord clamped 60 seconds after delivery of baby
  Interventions: Procedure: Umbilical cord clamping

INTERVENTIONS:
Procedure: Umbilical cord clamping — The umbilical cord will be clamped and cut after delivery, with timing as specified in each arm

SUMMARY:
The purpose of this research study is to find out how delaying cutting the umbilical cord until one minute after delivery of the baby during a cesarean impacts the amount of blood the mother loses during surgery. The study will also examine the benefits to the newborn from delayed cord clamping during cesarean.

DETAILED DESCRIPTION:
After delivery of a baby, the umbilical cord is cut to separate the baby from the placenta and the mother. The best time to cut the umbilical cord of full term babies is unknown. Traditionally, the umbilical cord is cut immediately at birth. There is however, continued blood flow from the placenta to the baby after delivery and so there may be a benefit to the baby from waiting to cut the cord until one minute after delivery. Studies show that delaying cutting the cord until at least one minute after delivery increases a full term baby's blood count in first two days of life and increases the baby's iron levels. The impact of delaying cutting the umbilical cord on a mother's health is not fully known. Delaying cutting the cord has minimal impact on the mother's health when the baby is delivered vaginally, but it is not known how delaying cutting the cord impacts the mother's health (and specifically the amount of blood a mother loses at delivery) when the baby is delivered by cesarean.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation
* Scheduled cesarean delivery at term (>=37 weeks)

Exclusion Criteria:

* Placenta previa
* Placenta abruption
* Intrauterine growth restriction with abnormal Dopplers
* Fetal anomalies
* Known fetal anemia
* Planned cord blood banking
* Preeclampsia
* Significant maternal anemia (Hgb <=7)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Maternal change in hemoglobin on post-operative day #1 | Baseline to postoperative day #1 (range 1-4 days)
  Difference in hemoglobin between routine pre-op CBC and a postpartum CBC collected on postoperative day #1, by venipuncture

SECONDARY OUTCOMES:
Postpartum hemorrhage | From day of surgery to postpartum discharge (average 3-4 days)
  Incidence of postpartum hemorrhage, defined as EBL >1000cc
Estimated blood loss | Day of surgery
  Estimated blood loss at cesarean delivery, based on estimation provider team
Need for Need for additional uterotonics | Day of surgery
  Administration of uterotonics (beyond standard pitocin) during cesarean
Maternal blood transfusion | From day of surgery to postpartum discharge (average 3-4 days)
  Transfusion of blood products during or after delivery
Venous cord blood Hgb/Hct | Day of delivery
  Obtained from cord blood sample
Neonatal Hgb/Hct | Day 0-2 of life
  Obtained from neonatal heel stick
APGAR scores | Day of delivery
  Assigned at delivery
Need for phototherapy for jaundice | From birth to hospital discharge (average 3-4 days)
  Any use of phototherapy

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Gyamfi-Bannerman, MD, Study Chair — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Purisch SE, Ananth CV, Arditi B, Mauney L, Ajemian B, Heiderich A, Leone T, Gyamfi-Bannerman C. Effect of Delayed vs Immediate Umbilical Cord Clamping on Maternal Blood Loss in Term Cesarean Delivery: A Randomized Clinical Trial. JAMA. 2019 Nov 19;322(19):1869-1876. doi: 10.1001/jama.2019.15995. PMID 31742629